CLINICAL TRIAL: NCT01001767
Title: Prospective Randomized Placebo Controlled Trial of Omega-3 Fatty Acids in HIV Infected Subjects to Modulate Cardiovascular Risk
Brief Title: Pilot Placebo Controlled Study With Lovaza in Cardiovascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: The Campbell Foundation (Other); Case Western Reserve University (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Grace McComsey, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AIDS 10-08-24
Record Dates: First submitted 2009-10-22; First posted 2009-10-27 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: HIV Infections; Heart Disease
Keywords: Omega-3 Fatty Acids; HIV; Heart Disease; Treatment experienced
MeSH Terms: conditions — HIV Infections; Heart Diseases | interventions — Omacor; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lovaza (Active Comparator): Lovaza 1 gram by mouth twice a day for 24 weeks.
  Interventions: Drug: Lovaza
- Placebo (Placebo Comparator): Placebo capsule by mouth twice a day x 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovaza — Lovaza one gram twice a day for 24 weeks
  Other Names: Omega-3 fatty acid
  Arms: Lovaza
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Several studies have shown that there is an increased risk of heart disease in people with HIV. In this study the investigators are looking at the effect of Lovaza (Omega-3 fatty acid) on improving endothelial function and decreasing inflammation which may contribute to this increased risk. The investigators will also be doing studies to analyze coagulation and inflammation markers.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Ages 18-70
* HIV-1 RNA <400 copies/ml.
* On stable ART (antiretroviral therapy) regimen for 12 weeks with no intent of modifying regimen, and cumulative ART before study entry of 12 mos.

Exclusion Criteria:

* Active infection
* Inflammation or malignancy
* Uncontrolled diabetes or hypothyroidism
* LDL (low density lipoprotein) cholesterol >160 and triglyceride levels >750
* Framingham risk score <6.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Hileman CO, Carman TL, Storer NJ, Labbato DE, White CA, McComsey GA. Omega-3 fatty acids do not improve endothelial function in virologically suppressed HIV-infected men: a randomized placebo-controlled trial. AIDS Res Hum Retroviruses. 2012 Jul;28(7):649-55. doi: 10.1089/aid.2011.0088. Epub 2011 Oct 17. PMID 21870979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 22, 2009 to September 1, 2009 35 individuals were enrolled and randomized. Participants were recruited from the Special Immunology Unit at University Hospitals Case Medical Center and from other HIV clinics in Cleveland, Ohio.
Pre-assignment Details: No wash out, run-in or transition period required for this study.
Groups:
- Lovaza: Lovaza 1 gram by mouth twice a day x 24 weeks
Period: Overall Study
Arm/Group | Lovaza | Placebo
Started | 18 | 17
Completed | 14 | 17
Not Completed | 4 | 0
Not completed — no baseline study performed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lovaza | Placebo | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [47 to 53] | 51 [49 to 54] | 51 [48 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 17 | 35
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow Mediated Dilation (FMD) of the Brachial Artery
Description: Flow mediated dilation (FMD) of the brachial artery measured by ultrasound is a measure of endothelium dependent endothelial cell function. FMD is expressed as a percent change from baseline brachial artery diameter to brachial artery diameter after reactive hyperemia.
Time Frame: baseline and week 24
Population: Randomized to have equal number in both groups
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 14 | 17
percent change | -0.13 (2.60) | 1.47 (4.05)

ADVERSE EVENTS:
Arm/Group | Lovaza | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

LIMITATIONS AND CAVEATS:
Small sample size may have precluded our ability to detect a small effect. Pill counts were used to monitor adherence. All participants were male.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No